CLINICAL TRIAL: NCT06862531
Title: COVERT : A Single-center, Interventional Diagnostic Study With Minimal Risks and Constraints, Aimed at Longitudinally Evaluating Serum Antibody Levels in Patients With COVID-19 According to the Severity of Their Symptoms.
Brief Title: A Single-center, Interventional Diagnostic Study With Minimal Risks and Constraints, Aimed at Longitudinally Evaluating Serum Antibody Levels in Patients With COVID-19 According to the Severity of Their Symptoms.
Acronym: COVERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioaster (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A02008-31
Record Dates: First submitted 2025-03-05; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe (Other): patients who developed a severe form of Covid (hospitalized in ICU in March/April 2020)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — A sample of blood (1mL) was taken

SUMMARY:
The COVERT protocol was designed to assess, through a longitudinal analysis, the level of antibodies present in the serum of patients with COVID-19, the duration and the persistence of the humoral response in correlation with the severity of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old,
* Patient whose Covid-19 diagnosis has been confirmed by RT-PCR test (SARS-CoV-2 positive) from a nasopharyngeal swab/broncho alveolar lavage
* Patient whose severity of Covid-19 required hospital treatment
* Patient whose Covid-19 form is defined as moderate (stay in general ward) or severe (stay in ICU), based on the clinical evaluation conducted by the doctor
* Patient agreeing to participate in the study and having signed the informed consent.

Exclusion Criteria:

* Adult person subject to legal protection,
* Pregnant, parturient or breastfeeding woman
* Person not affiliated to a social security scheme or not beneficiary of such a scheme
* Person subject to a safeguard measure
* Person deprived of liberty by a judicial or administrative decision and woman hospitalized without consent under Articles L.3212-1 and 3213-1, which do not fall under Article L.1122-8 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
The correlation between serum antibody levels (IgM/IgG), the stage of the disease (in relation to the onset date of symptoms), and the severity of the disease (severe form versus moderate form) | 10month after inclusion
  The correlation between serum antibody levels (IgM/IgG), the stage of the disease (in relation to the onset date of symptoms), and the severity of the disease (severe form versus moderate form)

CONTACTS AND LOCATIONS:
Locations (1):
- CH ANnecy-GEnevois (CHANGE), Metz-Tessy, Auvergne-Rhône-Alpes, France